CLINICAL TRIAL: NCT05214300
Title: Screening for Bleeding Disorders in Children: Evaluation of the Elements of the Interrogation, the Screening Workup and the Clinical Scores
Brief Title: Screening for Bleeding Disorders in Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0648
Record Dates: First submitted 2021-12-24; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-12

CONDITIONS: Bleeding Disorder
Keywords: von Willebrand disease; hemophilia A and B; other coagulant factor deficiencies
MeSH Terms: conditions — Hemostatic Disorders; von Willebrand Diseases; Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators try to improve the screening of bleeding disorders in children by identifying symptoms, laboratory abnormalities and clinical scores discriminating patients congenital bleeding disorders in order to create a simple screening algorithm applicable in pediatrics, aiming for use in pre-anesthetic consultation and in consultation by pediatricians and general practitioners.

DETAILED DESCRIPTION:
Objective : To determine simple clinical and biological factors that can improve the screening of hemostatic diseases at risk of hemorrhage in children.

Method:

* Retrospective inclusion of all patients <18 years referred to the CRTH in pediatric consultation for the reason of exploration of a hemorrhagic syndrome or exploration of an anomaly in the hemostasis assessment.
* Data collected (by collection in the medical file):

Patient data: Age, sex, personal and family history of hemorrhagic disease

Clinical data: hemorrhagic symptomatology (epistaxis, gingivorrhagia, etc.) Biological data: PT, TCK, factor assay, platelet function Medical data: complete diagnosis if diagnosis of hemorrhagic disease

* Scores: HEMOSTOP, PBQ, ISTH, TOSETTO score
* Analyzes: calculation of the Odd Ratio, AUC, Se, Sp, VPP, VPN for different clinical / biological factors and each score.

ELIGIBILITY:
Inclusion criteria:

* referred by their general practitioner or another caring physician for evaluation of bleeding symptoms
* abnormal laboratory test results or family study
* the patient being the first-degree relative of a patient with a known bleeding disorder.

Exclusion criteria:

- older than 18 years old.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children 0-18 years old
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Observe the correlation between the data of the interrogation | 1 day
  Observe the correlation between the data of the interrogation, the clinical examination and the clinical history and the demonstration of a confirm congenital bleeding disorder.

OTHER OUTCOMES:
Test scores | day 1
  Test scores (HEMOSTOP, TOSETO ...) to propose a simple algorithm for carrying out screening assessments for congenital bleeding disorders in children.
Compare several scores | day 1
  Compare several scores (HEMOSTOP, TOSETO ...) to propose a simple algorithm for carrying out screening assessments for congenital bleeding disorders in children.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre THERON, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC